CLINICAL TRIAL: NCT04708574
Title: Impact of Lifestyle Changes on Reducing Risk Factors for Type 2 Diabetes Among Arab Canadian Muslim Women.
Brief Title: Lifestyle Changes Reducing Type 2 Diabetes Risk Among Arab Canadian Muslim Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Michelle Mottola, Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12132E
Record Dates: First submitted 2021-01-08; First posted 2021-01-14 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Lifestyle Risk Reduction; Type2 Diabetes
Keywords: type 2 diabetes; risk reduction; lifestyle intervention; Arab Canadian Muslim women
MeSH Terms: conditions — Risk Reduction Behavior; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group attended a supervised exercise program for women only that presented Arabic music and traditional dance steps (the Lebanese Dabka) three times a week in the London Muslim Mosque Gym. The intervention lasted 12 weeks. There was also a nutrition education component that occurred once per week for the duration of the intervention. The lifestyle intervention group was instructed to walk 10,000 steps per day for the 12 weeks of the program. They were given instructions to take a 30-min walk on days when no formal exercise sessions were offered.
  Interventions: Behavioral: Lifestyle intervention
- Control (Placebo Comparator): The control group participants followed their typical work and leisure routines during the weeks of investigation. The women in the control group were offered the same intervention at the end of the 12 weeks.
  Interventions: Other: Placebo - Control

INTERVENTIONS:
Behavioral: Lifestyle intervention
  Arms: Intervention
Other: Placebo - Control
  Arms: Control

SUMMARY:
Aim: The purpose was to investigate whether modifiable risk factors for type 2 diabetes can be reduced by an intensive healthy lifestyle intervention designed for Arab Muslim women.

Methods: Women were assigned randomly to either an Exercise and Nutrition Group (ENG) or a Control Group (CG). The ENG attended a women-only supervised exercise program that presented Arabic music and traditional Lebanese Dabka steps three times/week in the Mosque Gym for 12 weeks. A nutritionist was available one hour/week for nutrition education. The CG followed their typical day.

DETAILED DESCRIPTION:
Women were assigned randomly using a computer-generated random numbers table to either an Exercise and Nutrition Group (ENG) or a Control Group (CG). The women received step-by-step instructions on how to complete a consecutive 3-day food record (including two week-days and one weekend day) and an exercise log for 7 days using a pedometer (YAMAX SW-200 Digi-Walker) to determine steps/day. The information and instruction were delivered to the women in English or Arabic. Body weight and height were measured to the nearest 0.1 kg and 0.1 cm, respectively. Women came to the lab after a 12 hour fast and a blood sample was drawn. Waist and hip measurements were taken along with resting blood pressure. Estimated fitness levels was measured by a trained kinesiologist using a Step Test (Siconolfi et al. 1985). All baseline measurements, including the 3-day food intake record and the 7-day pedometer step count log were repeated at the end of the 12-week intervention in both groups. The ENG group attended a supervised women-only exercise program that presented Arabic music and traditional dance steps (the Lebanese Dabka) three times a week in the London Muslim Mosque Gym and received nutrition education over the 12 weeks, one session per week.

ELIGIBILITY:
Inclusion Criteria:

* family history of type 2 diabetes (at least one parent),
* overweight or obese,
* been in Canada more than 10 years,
* mild hypertension,
* impaired glucose tolerance, or previous gestational diabetes (including giving birth to babies 4.0 kg or more),
* a sedentary lifestyle

Exclusion Criteria:

* uncontrolled hypertension,
* unstable angina,
* pulmonary and metabolic disease,
* severe arthritis or rheumatologic problems,
* already engaged in regular exercise training,
* pregnancy,
* menopause,
* already enrolled in a clinical research trial

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2006-03-08 (Actual); Primary Completion 2007-05-31 (Actual); Study Completion 2007-05-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline to post intervention for estimated fitness assessment test | Baseline and at the end of the 12 weeks
  Step test
Change in nutrition assessment from baseline to post intervention | Baseline and at the end of the 12 weeks
  From a 3-day food intake record

SECONDARY OUTCOMES:
Change in blood glucose values from baseline to post intervention | Baseline and at the end of the 12 weeks
  Fasted
Change in blood pressure (systolic and diastolic) values from baseline to post intervention | Baseline and at the end of the 12 weeks
  Seated
Change in waist to hip ratio from baseline to post intervention | Baseline and at the end of the 12 weeks
  Waist and hip measurements to calculate waist to hip ratio
Change in steps per day from baseline to post intervention | baseline (7 days) and at the end of the 12 weeks (7 days)
  pedometer

CONTACTS AND LOCATIONS:
Overall Officials: Michelle F Mottola, PhD, Principal Investigator — Western University, Canada
Locations (1):
- Exercise and Pregnancy Lab, 2245, 3-M Centre - University of Western Ontario, London, Ontario, Canada

REFERENCES:
- [Derived] Hussien S, McManus R, Prapavessis H, Sopper MM, Mottola MF. Effect of Lifestyle on Reducing Risk Factors for Type 2 Diabetes among Arab Canadian Muslim Women: A Randomized Control Trial. Med Sci Sports Exerc. 2024 Feb 1;56(2):249-256. doi: 10.1249/MSS.0000000000003311. Epub 2023 Oct 11. PMID 38214539